CLINICAL TRIAL: NCT03611673
Title: At-Home Olfactory Training With Essential-Oil Based Scents
Brief Title: At-Home Olfactory Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00141820
Record Dates: First submitted 2018-06-05; First posted 2018-08-02 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Olfactory Disorder
Keywords: sense of smell; smell test; at-home smell test; essential oil; olfactory loss
MeSH Terms: conditions — Anosmia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: 15 Scents (Experimental): Participants will be asked to inhale 15 different scents two times a day.
  Interventions: Other: Smell Test
- Group B: 4 Scents (Active Comparator): Participants will be asked to inhale 4 different scents two times a day.
  Interventions: Other: Smell Test

INTERVENTIONS:
Other: Smell Test — Oils are used for each of the different scents. Each scent will be put on an aromatherapy inhaling stick.

SUMMARY:
The purpose of this study is to determine the impact of a twice daily at-home olfactory training program with a twenty scent, essential oil-based smell test in patients with olfactory dysfunction.

DETAILED DESCRIPTION:
This study randomizes participants to receive either a four scent or fourteen scent olfactory retraining protocol. Baseline olfaction will be tested with a currently commercially available smell test as well as an essential oil based smell test. The protocol involves twice daily retraining where the participant inhales the scent and makes a mental note of what they should be smelling. The training period is six months total with a visit at 3 months to re-assess smell function as well as at six months.

ELIGIBILITY:
Inclusion Criteria:

* Have clinical olfactory dysfunction

Exclusion Criteria:

* Pregnant women
* Unable to perform routine follow-up
* Current participation in another clinical trial during this trial
* Patients with dementia, Alzheimer's disease, Parkinson's disease, or other neurocognitive disorders
* Diagnosis of other systemic conditions known to impact the sinonasal cavity such as Wegener's granulomatosis, Churg Strauss, and immunodeficiency
* Patients who are allergic to any of the smells or components of our olfactory testing
* Chronic rhinosinusitis, malignant tumors and/or oncologic therapies (radiation/chemotherapy)
* History of surgery on the nose or paranasal sinuses
* Patients using medications that may impact olfactory function (i.e. corticosteroids)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-06-02 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Change in ability to detect odorants - Sniffin' Sticks | Change from Baseline to Month 6
  Sniffin Sticks are a battery of 12 scents within a tube. The subject smells each scent and then chooses from 4 multiple choice options which is the scent they smelled. Increased number of correct responses indicates better sense of smell. 12/12 is the maximum score. 0/12 is the minimum score.
Change in ability to detect odorants - AROMA | Change from Baseline to Month 6
  AROMA is a essential oil based test. The subject is asked to respond if they detect a smell. If yes, they proceed to a 4 multiple choice items and select the item the smell. If no, they proceed to the next item. Higher number correct indicates better sense of smell. It consists of 13 odorants and 1 blank. Improved sense of smell would also increase the number of correctly identified odorants out of the 14 (including noting the 1 blank).

SECONDARY OUTCOMES:
Questionnaire of Olfactory Disorders-Negative Statements (QOD-NS) | Change from Baseline to Month 6
  The QOD-NS includes 17 statements that are graded on a scale from 0 to 3. Total score ranges from 0 to 51. Higher QOD-NS scores reflect better quality of life.
SF-12 (Short Form Health Survey) | Change from Baseline to Month 6
  SF-12 is a validated general measure of quality of life instrument that includes physical and mental scales. There are a total of 12 questions. Each aspect of the scale is weighted differently to yield a composite score. In general, a higher score is associated with better health.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Villwock, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States